CLINICAL TRIAL: NCT00108550
Title: Efficacy of Antidepressants in Chronic Back Pain
Brief Title: Chronic Low Back Pain Research Project
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLNA-013-04S; NCT01828450 (obsolete NCT alias)
Record Dates: First submitted 2005-04-15; First posted 2005-04-18 (Estimated); Results first posted 2014-02-10 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2013-12

CONDITIONS: Chronic Low Back Pain
Keywords: analgesia; antidepressant agents; back pain; pain
MeSH Terms: conditions — Agnosia; Back Pain; Pain | interventions — Gabapentin; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Gabapentin 300 mg orally three times daily up to a maximum of 1200 mg orally three times daily for 12 weeks
  Interventions: Drug: gabapentin
- 2 (Sham Comparator): Inert placebo capsules identical in size and shape to the experimental capsules, one to three capsules taken orally three times daily for 12 weeks
  Interventions: Drug: Inert placebo

INTERVENTIONS:
Drug: gabapentin — Gabapentin 300m on Day 1, with daily or weekly increase to 3600 mg (maximum) by mouth by Week 5 of the 12-week trial
  Other Names: Neurontin
  Arms: 1
Drug: Inert placebo — Inactive placebo capsule, one capsule on Day 1 with daily or weekly increase to 9 capsules daily by Week 5 of the 12-week trial
  Other Names: sugar pill
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether gabapentin is efficacious as an analgesic for chronic low back pain.

DETAILED DESCRIPTION:
Chronic low back pain (CLBP) is a major health problem for the VA, affecting up to 15% of all veterans. Nationally, its medical and disability costs exceed $50 billion annually. Despite its impact, relatively little research evaluates treatment for CLBP. Wide variation in patterns of care suggests uncertainty over effective therapy. Most chronic back cases are not surgical candidates. The mainstays of medical treatment have been non-steroidal anti-inflammatory drugs (NSAIDs), muscle relaxants, opioids, and antidepressants. Non-steroidal drugs and muscle relaxants are effective for acute but not for chronic back pain. Opioids may provide analgesia but safety limits their use. Tricyclic antidepressants provide modest pain relief, separate from effects on depression. But it is clear additional research is needed to develop more effective pharmacotherapy. One approach favored by many authorities is determining if agents effective for one type of chronic pain syndrome (e.g., diabetic neuropathy) can be generalized to other syndromes, like chronic back pain. Another is to identify effective drug combinations, based on selecting drugs with differing therapeutic mechanisms.

This research is a program of rigorous randomized clinical trials testing the efficacy of antidepressants for analgesia in chronic back pain. Because chronic pain is a complex disorder, the program features a multidisciplinary research team, involving specialists in psychiatry, orthopedic surgery, psychology, anesthesiology, clinical pharmacology, and biomathematics. The research has both pragmatic and explanatory aims. Our strategy has been to test antidepressants with differing, and selective properties in an attempt to isolate therapeutic mechanisms. Thus, we began with trials using selective norepinephrine reuptake inhibitors, and selective serotonin reuptake inhibitors (SSRIs), rather than those with dual noradrenergic and serotonergic effects (e.g., amitriptyline, imipramine). To ensure applicability of results, we have used rigorous diagnostic procedures to identify patients with chronic back pain due to degenerative disk disease. To enhance generalizability we recruit primary care patients rather than tertiary pain clinic samples. Patients without major depression are studied to examine analgesia separate from antidepressant effects. Secondary outcomes address function and life quality.

We have conducted three controlled trials using identical recruitment and assessment methodology. The first, comparing a noradrenergic antidepressant (nortriptyline) with placebo, indicated that the noradrenergic agent provided clinically relevant analgesia. The second was a head-to-head comparison of a selective noradrenergic agent (maprotiline) with a selective serotonin reuptake inhibitor (SSRI, paroxetine). The noradrenergic agent outperformed the SSRI, which was equivalent to placebo. To clarify these results we explored whether efficacy might be evident only at specific drug concentrations. Therefore, the third study, has a prospective concentration design comparing the most potent and selective noradrenergic antidepressant (desipramine) to the standard SSRI, fluoxetine. Subjects were randomized to placebo or predetermined concentration windows reflecting low, medium, and high exposure to study drugs and followed for 12 weeks. Interim analysis suggests that low concentration desipramine outperforms placebo (p<0.05). It is also superior to mid-concentration and high exposure desipramine--as well as all exposure levels of the SSRI, which are equivalent to placebo.

In sum, all three studies supported noradrenergic analgesia in CLBP, and the two studies that evaluated SSRIs failed to find analgesia. This suggests noradrenergic activity, perhaps within a therapeutic window, may be primarily responsible for back pain analgesia. These findings have led us away from studies proposing combining noradrenergic and serotonergic agents. An alternative approach which builds on these data, but first employs another class of agents, seems reasonable. This strategy is to assess if gabapentin, a calcium channel blocker agent with demonstrated efficacy in neuropathic pain, can be extended to chronic back pain.

We conducted a double-blind, randomized assignment, 12-week, placebo controlled clinical trial of the efficacy of gabapentin. Non-depressed chronic low back pain patients (N = 130) will be randomized to placebo or high dose gabapentin (3600 mg/day or maximum tolerable dose). Analysis was by intent to treat. The primary efficacy assessment is mean pain intensity (Descriptor Differential Scale, DDS) at exit. Secondary outcomes are function and life quality (Oswestry Disability Index, Short Form-36, Quality of Well-Being Scale). Safety evaluation includes rating adverse events (Scandinavian Society of Psychopharmacology Committee on Clinical Investiagations Side Effects Rating Scale, UKU), standardized physical examination, and clinical laboratory testing. Results could provide explanatory insight into mechanisms of back pain, and address the pragmatic clinical need by primary care providers and others for effective therapy.

ELIGIBILITY:
Inclusion Criteria:

* Must be resident of the county of San Diego, California
* Ages 21-70 inclusive
* Low back pain (T-6 or below, secondary to degenerative disk or degenerative joint disease) present "on a daily basis" for the previous 6 months or longer, of at least "moderate" intensity determined by Descriptor Differential Scale (DDS) > 7
* English-speaking, literate, able to understand the study and communicate with the study team
* Presently not a candidate for back surgery (one prior back surgery permitted if it was > 5 years ago and resulted in complete relief)
* Discontinued muscle relaxants, anticonvulsants, antidepressants, and opioids at least two weeks before screening and agree to discontinue throughout study (can remain on stable dose of NSAIDs)
* If female, not pregnant or lactating; agrees to use reliable contraception throughout the study, and has negative pregnancy test at screening
* Gives informed consent.

Exclusion Criteria:

* A major coexisting medical illness (e.g., diabetes, renal or hepatic disease, chronic obstructive pulmonary disease, cancer, or class III or IV organic heart disease) that might increase risks of gabapentin, or major surgical or non-surgical intervention for any disorder within the past 12 months, since rehabilitation from treatment may confound study outcomes
* Significant coexisting orthopedic or pain problems; sciatica (pain, weakness, or dysesthesia solely in distribution of a lumbar spinal nerve, with or without reflex change) or back pain due to other disorders (e.g., fibromyalgia, vertebral fracture, osteomyelitis, metastatic cancer, rheumatoid arthritis; spinal stenosis)
* Diagnostic and Statistical Manual (DSM)-IV diagnosis of alcohol or other substance abuse or dependence (within the previous 12 months or positive urine toxicology at screening), current major depression or dysthymia; or lifetime bipolar disorder (I or II) (excluded because gabapentin is antidepressive and antimanic); or major anxiety disorder (e.g., panic disorder; or psychosis; or lifetime presence of cognitive impairment disorder (e.g. dementia)
* History of multiple adverse drug reactions or known allergy to gabapentin
* Use of psychotropics (e.g., antidepressants, anxiolytics), which would need to be continued during the study, or other drugs or agents (i.e., herbal preparations) which might interact with the study drug
* Prior treatment with the study drug
* Use of systemic corticosteroids or corticosteroid injections within three months of screening; or concurrent behavioral therapies, chiropractic treatment, or transcutaneous electrical nerve stimulation unit
* Renal impairment (creatinine > 1.8 mg/dL)
* Hepatic impairment (bilirubin > 1.5 X upper normal limit, or aspartate aminotransferase (AST) or alanine transaminase (ALT) > 2 X upper normal limit)
* Hematologic abnormality (hemoglobin < 9.4 gm/dL; absolute white blood cell (WBC) count < 3000/mm3, platelets < 100,000
* Pregnancy
* Immunosuppression
* Use of experimental drugs or participation in other clinical trials

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2004-10; Primary Completion 2009-07 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph H. Atkinson, MD, Principal Investigator — VA San Diego Healthcare System, San Diego
Locations (1):
- VA San Diego Healthcare System, San Diego, San Diego, California, United States

REFERENCES:
- [Derived] Atkinson JH, Slater MA, Capparelli EV, Patel SM, Wolfson T, Gamst A, Abramson IS, Wallace MS, Funk SD, Rutledge TR, Wetherell JL, Matthews SC, Zisook S, Garfin SR. A randomized controlled trial of gabapentin for chronic low back pain with and without a radiating component. Pain. 2016 Jul;157(7):1499-1507. doi: 10.1097/j.pain.0000000000000554. PMID 26963844

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment were January 2005 to June 2009 by newsprint advertisements to the general community, by word-of-mouth, and posting of flyers at primary care clinics at two performance sites (VA San Diego Healthcare System and University of Califonia Medical Center, San Diego).
Groups:
- Gabapentin: gabapentin capsule 1200mg three times a day for 12 weeks
- Placebo: Inert placebo capsules, 3 capsules three times a day for 12 weeks
Period: Overall Study
Arm/Group | Gabapentin | Placebo
Started | 55 | 53
Completed | 39 | 37
Not Completed | 16 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gabapentin | Placebo | Total
Number analyzed (Participants) | 55 | 53 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.40 (8.88) | 54.62 (11.38) | 56.04 (10.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 23
  Male | 45 | 40 | 85
Region of Enrollment [Number; unit: participants]
  United States | 55 | 53 | 108

OUTCOME MEASURES:

1. Primary Outcome: Transformed Descriptor Differential Scale-Pain Intensity Scores Adjusted for Time
Description: Self-report measure of "current" pain intensity of chronic back pain. Participants rate pain on a 20 point scale as being greater or less intense relative to 12 adjectival descriptor word anchors (eg, greater or less than "faint," "moderate," "strong"). Scores range from 0 to 20 with higher scores indicating higher pain intensity. Prior to analysis an order-preserving mean-matching variance-stabilizing transformation was applied to this measure placing it on a continuous 0-1.5 scale. The single values reported below represent adjusted means of transformed pain intensity over all time points.
Time Frame: Baseline to Week 12 with Interim Measurement at Weeks 1, 2, 3, 4, 5, 7 and 9
Population: Analysis of all randomized participants receiving study drug
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Gabapentin
Number analyzed (Participants) | 53 | 55
units on a scale | 0.6683 [0.6145 to 0.7220] | 0.6988 [0.6463 to 0.7512]
Statistical Analysis 1: Comparison: Placebo vs Gabapentin; The null hypothesis was that Gabapentin is no better than placebo in reducing back pain. A mean-matching variance stabilizing transformation was applied to Descriptor Differential Scale Pain intensity (DDS) scores. Scores were modeled as a function of time (week) and group (gabapentin, placebo) in a mixed effects model. Random (subject-specific)intercept and slopes were fitted to the data. With alpha = .05 and N = 65 per group power is .8 to detect effect size =.4 standard deviations (SD); Test type: Superiority or Other; p = 0.4237, Mixed Models Analysis — There was no need for multiple comparisons adjustment for the primary outcome, since there was only one. However, secondary analyses were adjusted for multiple comparisons; Effect of covariates (age, gender, etc) was evaluated (modeled as fixed effects) in secondary analyses; Mean Difference (Final Values) = 0.0305, 95% CI 2-sided [-0.044 to 0.105], Standard Error of Mean 0.038 — The analysis was performed on transformed (rather than raw) Descriptor Differential Score Pain Intensity scores

2. Secondary Outcome: Roland and Morris Disability Index Scores Adjusted for Time
Description: This questionnaire measures disability in everyday function due to back pain. It is a 24-item checklist asking patients to endorse whether or not back pain limits activities they normally do (eg, "I stay at home most of the time because of my back"). Scores range from 0 to 24, with higher scores indicating greater disability in everyday function due to back pain. The single values reported below represent adjusted means of scores over all time points.
Time Frame: Baseline to Week 12 with Interim Measurement at Weeks 1, 2, 3, 4, 5, 7 and 9
Population: Randomized participants who received one dose of study drug
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Gabapentin
Number analyzed (Participants) | 53 | 55
units on a scale | 7.50 (4.30) [6.47 to 8.52] | 6.96 (3.53) [5.95 to 7.97]
Statistical Analysis 1: Comparison: Placebo vs Gabapentin; This is a secondary analysis; the null hypothesis is that Gabapentin performs no better than placebo in reducing the Roland and Morris score; Test type: Superiority or Other; p = 0.458, Mixed Models Analysis — Primary analyses was multivariable linear regression with fixed and random effects. After the Bonferroni adjustment a p-value would have been considered significant at 0.05 level if <0.01; Mean Difference (Final Values) = -.5343, 95% CI 2-sided [-1.940 to 0.872], Standard Error of Mean 0.7174

ADVERSE EVENTS:
Time Frame: Participant report of adverse effects at any point during the 12-week trial.
Description: A psychiatrist-administered, semi-structured interview (Scandinavian Society of Psychopharmacological Investigators Side Effect Rating Scale, UKU), assessed 48 psychotropic drug-associated symptoms in the prior 3 days. Items rated as "present" (of at least "mild" intensity) and "possibly" or "probably" drug-induced were counted as adverse effects.
Arm/Group | Placebo | Gabapentin
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/55
Other Adverse Events (participants affected / at risk) | 21/53 | 42/55
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=53) | Gabapentin (N=55)
sleepiness (Nervous system disorders) | 14 (14) | 29 (29)
asthenia/fatigue (Nervous system disorders) | 15 (15) | 27 (27)
orthostatic dizziness (Cardiac disorders) | 14 (14) | 24 (24)
decreased salivation (Gastrointestinal disorders) | 10 (10) | 22 (22)
increased sleep (Nervous system disorders) | 11 (11) | 21 (21)
concentration difficulties (Nervous system disorders) | 6 (6) | 21 (21)
accomodation disturbance (Eye disorders) | 3 (3) | 19 (19)
loss of balance (Nervous system disorders) | 2 (2) | 18 (18)
reduced sleep (Nervous system disorders) | 10 (10) | 7 (7)
constipation (Gastrointestinal disorders) | 9 (9) | 7 (7)
nausea (Gastrointestinal disorders) | 8 (8) | 7 (7)
polyuria/polydipsia (General disorders) | 6 (6) | 7 (7)
diarrhea (Gastrointestinal disorders) | 7 (7) | 6 (6)
increased dreaming (Nervous system disorders) | 5 (5) | 5 (5)
failing memory (Nervous system disorders) | 1 (1) | 9 (9)
erectile dysfunction (Reproductive system and breast disorders) | 2 (2) | 6 (6)
decreased sexual desire (Reproductive system and breast disorders) | 2 (2) | 5 (5)
weight gain (General disorders) | 1 (1) | 6 (6)
micturation disturbance (Renal and urinary disorders) | 4 (4) | 2 (2)
anxiety (Nervous system disorders) | 1 (1) | 5 (5)
headache (Nervous system disorders) | 2 (2) | 3 (3)
paresthesia (Nervous system disorders) | 3 (3) | 2 (2)

LIMITATIONS AND CAVEATS:
Limitations include small sample size, high rate of early termination, and moderate baseline levels of pain intensity and disability in everyday function which may have limited ability to detect an effect.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No